CLINICAL TRIAL: NCT01102699
Title: Bone Marrow Responsiveness to Pharmacologic Mobilization of Progenitor Cells in Diabetic Versus Non-diabetic Patients
Brief Title: Bone Marrow Progenitor Cell Mobilization in Diabetes
Acronym: GCSF-DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Angelo Avogaro, Professor of Endocrinology, University of Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GCSF-DM
Record Dates: First submitted 2010-04-09; First posted 2010-04-13 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; stem cells; bone marrow; mobilization
MeSH Terms: conditions — Diabetes Mellitus | interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Filgrastim, G-CSF (Experimental): Single s.c. dose of G-CSF (300 microg)
  Interventions: Drug: Filgrastim, hrG-CSF

INTERVENTIONS:
Drug: Filgrastim, hrG-CSF — Single subcutaneous injection of Filgrastim (hrG-CSF) 300 microg (30 MU)

SUMMARY:
Diabetes mellitus is associated with a significant reduction of circulating progenitor cells (CPCs). These include endothelial progenitor cells (EPCs), which are involved in cardiovascular homeostasis and repair. A reduction of CPCs in metabolic patients is associated with an increased risk of future adverse cardiovascular outcomes. Therefore, ways to active stimulate an increase of CPC levels in diabetes are actively pursued.

Experimental animal studies and preliminary data in humans indicate that a bone marrow defect is causally related to the low CPC level in diabetes.

Our previous data in rats indicate that diabetes reduces the bone marrow responsiveness to granulocyte colony-stimulating factor (G-CSF) in terms of progenitor cell mobilization.

In the present study, we aim at investigating bone marrow responsiveness to pharmacological mobilization of CPC in diabetic patients as compared to non-diabetic subjects.

DETAILED DESCRIPTION:
Diabetes mellitus is associated with a significant reduction of circulating progenitor cells (CPCs). CPCs are defined by the surface expression of the stem cell antigen CD34 and or CD133. These cells include endothelial progenitor cells (EPCs), which are involved in cardiovascular homeostasis and repair. EPCs are characterized by the co-expression of endothelial antigen(s), such as KDR.

A reduction of CPCs in metabolic patients is associated with an increased risk of future adverse cardiovascular outcomes, such as myocardial infarction, stroke, revascularization, etc. Therefore, ways to active stimulate an increase of CPC levels in diabetes are actively pursued. Indeed, there are several drugs that stimulate CPCs or EPCs, but it is not fully clear if they are active also in diabetic patients.

The mechanisms that account for CPC reduction in diabetes include defective bone marrow mobilization, reduced survival and increased homing outside the bloodstream. Experimental animal studies and preliminary data in humans indicate that a bone marrow defect is causally related to the low CPC level in diabetes.

Our previous data in rats indicate that diabetes reduces the bone marrow responsiveness to G-CSF in terms of c-kit+/Sca-1+ progenitor cell mobilization.

There is also some experimental evidence in type 2 diabetic rats that a specific form of autonomic neuropathy impairs bone marrow mobilization of progenitor cells.

In the present study, we aim at investigating bone marrow responsiveness to pharmacological mobilization of CPC in diabetic patients as compared to non-diabetic subjects.

Diabetic subjects and control subjects will be administered with a single dose of granulocyte colony stimulating factor (G-CSF) and progenitor cells will be quantified before and 24 hours after G-CSF administration. Progenitor cells will be analyzed by flow cytometry on the basis of the expression of CD34, CD133 and KDR.

Mean percentage variation of CPCs and EPCs will be compared in diabetic versus non diabetic patients to understand whether or not diabetes is associated with a significant defective mobilization of progenitor cells.

As a secondary aim, diabetic patients will be divided in those with and without diabetic autonomic neuropathy (DAN) to understand if DAN modulates bone marrow responsiveness to G-CSF.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus (for cases) or absence of diabetes (for controls);
* Age 25-65;
* Both sexes;
* Capability of providing informed consent.

Exclusion Criteria:

* Age <25 or >65;
* Fertile women;
* Recent (within 2 months) acute illnesses;
* Chronic immune of infectious diseases;
* Current or remote hematological disorders;
* Leukocytosis, leukopenia or thrombocytopenia;
* Organ transplantation or immune suppression;
* Altered liver function;
* Severe renal failure (eGFR<30 mL/min/m2);
* Anomalies in lymphocytes subpopulations;
* High basal level of CD34+ cell count;
* Allergy to Filgrastim;
* Bronchial asthma or other chronic lung disorders;
* Current or remote cancer;
* Deny or impossibility to provide informed consent.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
CPC mobilization after a single G-CSF dose | 0-24 hours
  Circulating progenitor cell level will be assessed before and 24 hours after a single G-CSF dose in both diabetic and non diabetic patients.
  Change in CPC level will be indicative of bone marrow mobilization. Mobilization will be compared in diabetic versus non diabetic subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Avogaro, MD PhD, Principal Investigator — Dept. of Medicine, University of Padova, Medical School, Padova (Italy); Gian Paolo Fadini, MD, Study Director — Department of Medicine, University of Padova.
Locations (1):
- University Hospital, Division of Metabolic Diseases, Padua, Italy

REFERENCES:
- [Derived] Fadini GP, Albiero M, Vigili de Kreutzenberg S, Boscaro E, Cappellari R, Marescotti M, Poncina N, Agostini C, Avogaro A. Diabetes impairs stem cell and proangiogenic cell mobilization in humans. Diabetes Care. 2013 Apr;36(4):943-9. doi: 10.2337/dc12-1084. Epub 2012 Oct 30. PMID 23111057